CLINICAL TRIAL: NCT06358755
Title: Combination Effect of Optical Defocus and Low Dose Atropine in Myopia Control - a Randomized Clinical Trial
Brief Title: Combination Effect of Optical Defocus and Low Dose Atropine in Myopia Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10211476; P0041308 (Other: The Hong Kong Polytechnic University)
Record Dates: First submitted 2024-03-20; First posted 2024-04-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Myopia
Keywords: Myopia control; Defocus; Atropine
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated into 2 groups. One group will receive low dose atropine (0.01%) plus DIMS spectacles (ATD Group); another one will receive low dose atropine (0.01%) plus single vision spectacles (AT Group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, including ophthalmologists and optometrists, who are responsible for collection of data related to myopia progression and analysis of data will be blinded to study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose atropine plus DIMS (Experimental): This group will receive 0.01% atropine (twice per day: 1 drop in the morning and 1 drop at night before bedtime) and Defocus Incorporated Multiple Segments (DIMS) spectacle lenses
  Interventions: Device: Defocus Incorporated Multiple Segments lenses; Drug: Low dose atropine
- Low dose atropine (Experimental): This group will receive 0.01% atropine (twice per day: 1 drop in the morning and 1 drop at night before bedtime) and single vision spectacle lenses
  Interventions: Device: single vision spectacle lenses; Drug: Low dose atropine

INTERVENTIONS:
Device: Defocus Incorporated Multiple Segments lenses — Defocus Incorporated Multiple Segments lenses that provide optical defocus for myopia control will be given to this group of participants.
  Arms: Low dose atropine plus DIMS
Device: single vision spectacle lenses — Single vision spectacle lenses will be given to this group of participants.
  Arms: Low dose atropine
Drug: Low dose atropine — 0.01% atropine administrated twice per day (1 drop in the morning and 1 drop at night before bedtime) will be given as intervention.

SUMMARY:
The purpose of the study is to investigate the combination effect of optical defocus and low dose atropine on myopia control in schoolchildren.

DETAILED DESCRIPTION:
This study is a two-arm randomised controlled trial with a 18-month duration. Participants will be healthy Hong Kong Chinese schoolchildren with low to moderate myopia. The aim is to determine the combination effect of optical defocus and low dose atropine on myopia control in schoolchildren. Optical defocus will be delivered by Defocus Incorporated Multiple Segments (DIMS) spectacle lenses.

A total of 112 Hong Kong Chinese children aged 7 to 12 years (56 in each group) will be recruited and randomly allocated into two groups. One group will receive low dose atropine (0.01%) plus DIMS spectacles (ATD Group); another one will receive low dose atropine (0.01%) plus single vision spectacles (AT Group).

They must have no prior or current myopia control treatment, have no ocular or systemic diseases/abnormalities that affect visual function, refractive development or spectacle lens wear, and no previous intraocular or corneal surgery. They must not have allergy to atropine.

Their cycloplegic refraction and axial length will be monitored every six months for 18 months. The changes in refractive errors and axial length between groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment: 7 to 12 years
* Ethnicity: Hong Kong Chinese
* Myopia: -0.75D (in spherical equivalent) or above in both eyes
* Astigmatism: -1.50D or less in both eyes
* Anisometropia: 1.50D or less (in spherical equivalent) between two eyes
* Best corrected monocular visual acuity (VA): 0.04 logMAR or better
* Ocular health: No abnormalities in both internal and external ocular health
* Systemic health: No abnormalities such as cardiac and respiratory diseases
* Binocular vision: No strabismus, diplopia, suppression and other binocular abnormalities
* Normal colour vision
* No previous refractive surgery or use of myopic control interventions, such as atropine, orthokeratology, and specialized spectacle lenses and contact lenses for myopic control
* Able to wear the prescribed spectacles
* No known allergy to atropine

Exclusion Criteria:

* Eye disease or binocular vision problems (e.g., strabismus, amblyopia, oculomotor nerve palsies, corneal disease, etc.)
* Previous intraocular or corneal surgery
* Colour vision deficiencies
* Systemic disease that may affect vision, vision development (e.g. diabetes mellitus, hypertension, Down syndrome, etc.)
* Systemic disease that are contradictory to atropine (e.g. asthma, cardiac diseases, etc.)
* Previous gas permeable, soft bifocal, or orthokeratology contact lenses wear or bifocal / progressive addition lens spectacles wear or use of atropine or pirenzepine (longer than one month of usage)
* Previous or current participation in myopia control studies
* Allergy to cyclopentolate hydrochloride or atropine

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cycloplegic refraction | Baseline, 6th month, 12th month and 18th month
  Changes in cycloplegic refraction in spherical equivalent (Dioptres) over 18 months from baseline will be measured.
Changes in axial length | Baseline, 6th month, 12th month and 18th month
  Changes in axial length (mm) over 18 months from baseline will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ka Man Chun, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Centre for Myopia Research, The Hong Kong Polytechnic University and Department of Ophthalmology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chun RKM, Hon Y, Law TK, Wong KYQ, To CH, Shih KC, Leung CKS, Tse DYY. Combination effect of optical defocus and low dose atropine in myopia control: Study protocol for a randomized clinical trial. PLoS One. 2024 Jun 26;19(6):e0306050. doi: 10.1371/journal.pone.0306050. eCollection 2024. PMID 38923965